CLINICAL TRIAL: NCT01343758
Title: A Double-blind Randomized Controlled Clinical Trial Investigating the Use of Intravenous Dextrose for Dehydration and Ketosis in Children With Gastroenteritis and Dehydration.
Brief Title: Study Investigating the Use of Intravenous Fluids With Dextrose for Dehydrated Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Jason Levy (PI), Children's Hospital Boston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-11-153
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Gastroenteritis; Dehydration
MeSH Terms: conditions — Gastroenteritis; Dehydration | interventions — Glucose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5% dextrose in normal saline (Active Comparator): This group will receive a bolus of normal saline that contains 5% dextrose
  Interventions: Other: 5% dextrose in normal saline
- Normal Saline Bolus (No Intervention)

INTERVENTIONS:
Other: 5% dextrose in normal saline — Subjects will be randomized to receive a intravenous fluid bolus of 5% dextrose in normal saline or normal saline
  Arms: 5% dextrose in normal saline

SUMMARY:
Infants and young children often become infected with gastroenteritis leading to vomiting and diarrhea. This can lead to dehydration, one of the most common complaints in the Pediatric Emergency Department. These children are often in need of treatment with intravenous (IV) fluids. While the investigators know that IV fluids work, it is not clear which type or how much fluid is the best amount to give. Currently, the most common type of IV fluid given is salt water, also called normal saline.

In contrast to adults, infants and young children with dehydration often have a build up of a certain type of acid in their blood which can perpetuate the nausea, vomiting, and general malaise associated with gastroenteritis. The investigators feel that giving these children IV fluids with lots of sugar (in addition to the salt) reduces the acid more rapidly than giving just salt water alone. In a prior study, the investigators have shown that children who receive lower amounts of sugar in the IV fluids return to the Emergency Department more often for a second visit. Based on this study, the investigators believe that children who receive the sugar-salt solution will do better than children who receive just normal saline.

The investigators will determine if the sugar-salt solution is better by giving equal numbers of children the sugar-salt solution and normal saline and then see what happens to each child. The investigators will monitor who needs to be admitted, how much each child vomits, how much each child drinks, and also the level of acid in the blood before and after getting the IV fluid. After the study is completed, the investigators can compare the two different groups (children who received the sugar-salt solution versus children who received normal saline alone) to determine if one group had greater improvement and better clinical outcome than the other.

ELIGIBILITY:
Inclusion Criteria:

* 6 months to 6 years of age
* Gastroenteritis
* Requires IV fluids for dehydration

Exclusion Criteria:

* Chronic disease
* Comorbid condition
* Received IV fluids or antiemetics in the last 12 hours
* Symptoms for more than 7 days
* Blood glucose less than 40

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 188 (Estimated)
Dates: Start 2007-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Admission Rate | During emergency department visit
  The investigators will measure what percentage of patients in each treatment group are admitted.

SECONDARY OUTCOMES:
Change in Serum Ketones | 1 and 2 hours after treatment given
  The investigators will measure the change in serum ketones at 1 and 2 hours after the study fluid is given and compare the mean change in each treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Levy, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States